CLINICAL TRIAL: NCT05146778
Title: A Single-blinded Randomized-controlled Study to Reduce Persistent Post-mastectomy Pain Using Multimodal Opioid-free Anesthesia
Brief Title: A Study to Reduce Persistent Post-mastectomy Pain Using Opioid-free Anesthesia
Acronym: RELIEF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Sung Gwe Ahn, Assocaite Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-0568-001
Record Dates: First submitted 2021-09-23; First posted 2021-12-07 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Mastectomy; Pain, Chronic; Pain, Post Operative
MeSH Terms: conditions — Breast Neoplasms; Chronic Pain; Pain, Postoperative | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: 1. Control arm: Conventional Anesthesia with opioid
  2. Interventional arm: Opiod-free Anesthesia with dexmedetomidine and lidocaine
Who Masked: Participant
Masking Description: Patients will be not aware of which type of anesthesia would be applied during operation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid-free anesthesia group (Active Comparator): OFA group will be sedated using dexmedetomidine and lidocaine during mastectomy.
  Interventions: Procedure: Opioid-free anesthesia
- Conventional anesthesia group with opioid (Active Comparator): Conventional opioid anesthesia group will be sedated using remi-fentanyl during mastectomy.
  Interventions: Procedure: Conventional opioid-based anesthesia

INTERVENTIONS:
Procedure: Opioid-free anesthesia — OFA group will be sedated using dexmedetomidine and lidocaine.
  Other Names: Dexmedetomidine and lidocaine-based anesthesia
  Arms: Opioid-free anesthesia group
Procedure: Conventional opioid-based anesthesia — Conventional opioid-based anesthesia group will be sedated using remi-fentanyl
  Other Names: Remi-fentanyl
  Arms: Conventional anesthesia group with opioid

SUMMARY:
In 230 patients undergoing mastectomy, the investigators will compare opioid-free anesthesia (OFA) versus conventional opioid-based anesthesia in terms of chronic pain. The enrolled patients will be randomly assigned into two groups with 1:1 ratio. Chronic pain will be evaluated at 1 year after mastectomy based on the Breast Cancer Pain Questionnaire (BCPQ). Baseline pain sensitivity test and psychologic evaluation will be done before operation.

DETAILED DESCRIPTION:
Study population

1. All of patients will undergo mastectomy with or without immediate breast reconstruction.
2. 230 patients will be enrolled.

Intervention

1. OFA group will be sedated using dexmedetomidine and lidocaine.
2. Conventional opioid anesthesia group will be sedated using remifentanil.

Pain screening

1. Breast Cancer Pain Questionnaire (BCPQ)
2. Pain-detect, HADS, EQ-5D, PHQ-15 (somatic symptom), PCS (pain catastrophizing), BFI (big five inventory), HAM-A&D, Pressure algometry (Pain sensitivity), Quantitative sensory test (pinprick)

ELIGIBILITY:
Inclusion Criteria:

* All of patients will undergo mastectomy with or without immediate breast reconstruction.

Exclusion Criteria:

* Previous history of breast surgery
* Allergy to drug
* Other cancer history
* Underlying psychologic disorder
* Patients with chronic pain requiring pain killers
* Baseline SpO2 <95%
* Left ventricular EF <40%
* Bradycardia as HR <50 bpm
* BMI >35kg/m2
* Pregnant woman

Ages: 19 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2021-12-16 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
chronic breast pain at 1 year after mastectomy | 1 year after mastectomy
  chronic pain will be assessed by Breast Cancer Pain Questionnaire (BCPQ). Zero score means absence of persisting breast-related pain. The minimum and maximum values of pain scale are 0 and 11, respectively. High score means worse outcome. Moderating role of preoperative psychosocial factors on the impact of OFA on chronic postoperative pain will be evaluated.

SECONDARY OUTCOMES:
psychological symptoms | 1 year after mastectomy
  Presence of anxiety and depression symptoms will be assessed by HADS (Hospital Anxiety and Depression Scale) questionnaire. The range of each symptoms scale is between 0 and 21. A scale of 0-7 is defined as normal, a scale of 8-10 is defined as borderline, and a scale of 11-21 is defined as abnormal. High score means worse outcome.
Pain Sensitivity | 1 year after mastectomy
  The type of pain will be assessed by painDetect Questionnaire (PDQ). The PDQ comprises 12 items. The first three assess current pain, strongest pain during the past 4 weeks, and average pain during the past 4 weeks on a 0-10 point numerical rating scale from "none" to "worst imaginable".

CONTACTS AND LOCATIONS:
Overall Officials: Sung Gwe G Ahn, M.D.,Ph.D., Principal Investigator — Gangnam Severance Hospital
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No